CLINICAL TRIAL: NCT02991703
Title: Simplified Pulse Wave Velocity Measurement, Validation Study of the pOpmètre in Children
Acronym: EPIPOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC16_0161
Record Dates: First submitted 2016-11-23; First posted 2016-12-13 (Estimated); Last update posted 2024-05-13 (Actual); Status verified 2018-05

CONDITIONS: Cardiovascular Diseases; Arteriosclerosis; Atherosclerosis
Keywords: Arterial stiffness; pulse wave velocity; Sphygmocor; applanation tonometry; pOpmètre; children; EPIPAGE cohort
MeSH Terms: conditions — Cardiovascular Diseases; Arteriosclerosis; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SphygmoCor® (Active Comparator)
  Interventions: Device: Sphygmocor
- pOpmètre® (Experimental)
  Interventions: Device: pOpmètre®

INTERVENTIONS:
Device: pOpmètre® — the pOpmètre® uses saturation sensors,
  Arms: pOpmètre®
Device: Sphygmocor — the Sphygmocor uses applanation tonometry
  Arms: SphygmoCor®

SUMMARY:
Arterial stiffness is an important marker of cardiovascular risk. It is measured by pulse wave velocity. The reference device to measure pulse wave velocity is the Sphygmocor which uses applanation tonometry. It is used in adults and children. An easier method called pOpmètre using saturation sensors is validated in adults but not in children. The objective of this study is to compare the pulse wave velocity values measured with the pOpmètre® with those of the SphygmoCor® to validate the pOpmètre in children between 4 and 8 years old.

DETAILED DESCRIPTION:
Prematurity is associated with an increased risk of developing cardio-vascular diseases in adulthood : a low birth weight linked to prematurity is correlated to a higher coronary disease mortality rate, a higher blood pressure level in adulthood, to abnormal glucose metabolism regulation, and to signs of nephron reduction. An independent marker of cardiovascular risk is arterial stiffness: it is associated with a higher risk of major cardiovascular events including stroke, acute coronary syndrome and complications of end-stage renal disease. It is measured by pulse wave velocity which is the gold standard in adulthood. Pulse wave velocity is also correlated to cardiovascular risk in childhood. National cohort EPIPAGE II is made of 4290 premature babies born in 2011. A study is scheduled at 5 years old and a half including a medical examination and a neuropsychological evaluation. An ancillary study lengthening medical consultation for 15 minutes is scheduled with 750 to 1000 of these children for a more precise vascular evaluation including pulse wave velocity. Different methods can be used to measure pulse wave velocity in children: these include applanation tonometry devices such as the SphygmoCor ® system. Its reference values are well known in adulthood and were determined more recently in childhood. It is the reference device but it is expensive, can be used only in expert health centres and time of measurement is long. In children, an easier-to-use and faster device would be more advantageous. The pOpmètre® uses 2 distal oxygen saturation sensors on finger and toe to deduce pulse wave velocity. This device has already been validated in adults. The aim of this study is to validate the pOpmètre in children between 4 and 8 years old. In that purpose, patients are installed in the supine position, at rest. The child's mensurations are measured. The two pOpmètre sensors are put on finger and toe. Blood pressure is measured by an armband on the right limb. Then another armband is put around the thigh and a tonometer is applied on the right carotid which allows pulse wave velocity measuring by the Sphygmocor. Pulse wave velocity is measured with the pOpmètre using the time delay between finger pulse signal and toe pulse signal. The values got with the two devices are compared using a Bland and Altman graph. The pOpmètre is considered to be validated if the 95% confidence interval of the bias is included between -0.5 m/sec and 0.5 m/sec that is about 10% of the normal value at that age (5.0 m/s +/-0.13).

ELIGIBILITY:
Inclusion Criteria:

* children between 4 and 8 years old hospitalized in the Mother and Children Hospital in Nantes during the study period.

Exclusion Criteria:

* Vasoconstrictor treatment,
* compressive bandage on the measured area,
* peripheral venous access on the measured side,
* vascular surgery or pathology on the measured area,
* significant pain or agitation,
* parental or legal representative disapproval,
* child disapproval.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Difference between the two simultaneous measurements of velocity of the pulse wave by the pOpmeter® and the Sphygmocor®. | Day One

REFERENCES:
- [Background] Willum-Hansen T, Staessen JA, Torp-Pedersen C, Rasmussen S, Thijs L, Ibsen H, Jeppesen J. Prognostic value of aortic pulse wave velocity as index of arterial stiffness in the general population. Circulation. 2006 Feb 7;113(5):664-70. doi: 10.1161/CIRCULATIONAHA.105.579342. PMID 16461839
- [Background] Urbina EM, Williams RV, Alpert BS, Collins RT, Daniels SR, Hayman L, Jacobson M, Mahoney L, Mietus-Snyder M, Rocchini A, Steinberger J, McCrindle B; American Heart Association Atherosclerosis, Hypertension, and Obesity in Youth Committee of the Council on Cardiovascular Disease in the Young. Noninvasive assessment of subclinical atherosclerosis in children and adolescents: recommendations for standard assessment for clinical research: a scientific statement from the American Heart Association. Hypertension. 2009 Nov;54(5):919-50. doi: 10.1161/HYPERTENSIONAHA.109.192639. Epub 2009 Sep 3. PMID 19729599
- [Background] Ancel PY, Goffinet F; EPIPAGE 2 Writing Group. EPIPAGE 2: a preterm birth cohort in France in 2011. BMC Pediatr. 2014 Apr 9;14:97. doi: 10.1186/1471-2431-14-97. PMID 24716860
- [Background] Reference Values for Arterial Stiffness' Collaboration. Determinants of pulse wave velocity in healthy people and in the presence of cardiovascular risk factors: 'establishing normal and reference values'. Eur Heart J. 2010 Oct;31(19):2338-50. doi: 10.1093/eurheartj/ehq165. Epub 2010 Jun 7. PMID 20530030
- [Background] Reusz GS, Cseprekal O, Temmar M, Kis E, Cherif AB, Thaleb A, Fekete A, Szabo AJ, Benetos A, Salvi P. Reference values of pulse wave velocity in healthy children and teenagers. Hypertension. 2010 Aug;56(2):217-24. doi: 10.1161/HYPERTENSIONAHA.110.152686. Epub 2010 Jun 21. PMID 20566959
- [Background] Curcio S, Garcia-Espinosa V, Arana M, Farro I, Chiesa P, Giachetto G, Zocalo Y, Bia D. Growing-Related Changes in Arterial Properties of Healthy Children, Adolescents, and Young Adults Nonexposed to Cardiovascular Risk Factors: Analysis of Gender-Related Differences. Int J Hypertens. 2016;2016:4982676. doi: 10.1155/2016/4982676. Epub 2016 Feb 18. PMID 26989504
- [Background] Alivon M, Vo-Duc Phuong T, Vignon V, Bozec E, Khettab H, Hanon O, Briet M, Halimi JM, Hallab M, Plichart M, Mohammedi K, Marre M, Boutouyrie P, Laurent S. A novel device for measuring arterial stiffness using finger-toe pulse wave velocity: Validation study of the pOpmetre(R). Arch Cardiovasc Dis. 2015 Apr;108(4):227-34. doi: 10.1016/j.acvd.2014.12.003. Epub 2015 Feb 11. PMID 25682547
- [Derived] Bichali S, Bruel A, Boivin M, Roussey G, Romefort B, Roze JC, Allain-Launay E. Simplified pulse wave velocity measurement in children: Is the pOpmetre valid? PLoS One. 2020 Mar 27;15(3):e0230817. doi: 10.1371/journal.pone.0230817. eCollection 2020. PMID 32218581
- See also: Related Info — https://www.youtube.com/watch?v=4aFnQ_0_bOI